CLINICAL TRIAL: NCT05809349
Title: The Mechanism of Theta Burst Stimulation (cTBS) in the Treatment of Drug-refractory Epilepsy Targeting the Dentate Nucleus of Cerebellum: An Exploratory Clinical Study
Brief Title: The Mechanism of cTBS Targeting Dentate Nucleus for DRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KY20232104
Record Dates: First submitted 2023-03-29; First posted 2023-04-12 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2023-03

CONDITIONS: Transcranial Magnetic Stimulation; Drug Resistant Epilepsy; Cerebellum
MeSH Terms: conditions — Drug Resistant Epilepsy | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DRE patients (Experimental): There will be 50 drug-refractory epilepsy (DRE) patients in this study.
  Interventions: Device: transcranial magnetic stimulation

INTERVENTIONS:
Device: transcranial magnetic stimulation — The stimulation intensity will be 80% resting motor threshold (RMT). The theta burst stimulation (cTBS) with a frequency at 50Hz, repeated at 5Hz, are delivered in a duration of 33.2s with the number of stimulation pulses of 600. Two groups of stimulation will be repeated in each cerebellar dentate nucleus with an interval of 5 min in each group. The treatment will last for 2 weeks, with 5 times per week.

SUMMARY:
In our previous cross-over study--the continuous θ burst stimulation (cTBS) targeting cerebellum dentate nucleus of 44 drug-refractory epilepsy (DRE) patients, a significant reduction in seizure frequency was observed. However, the mechanism of this target to reduce seizures is still unknown. This study aims to explore the mechanism of cTBS targeting cerebellum dentate nucleus for DRE, in order to provide theoretical support for this treatment method. A total of 50 patients with DRE will have 2-week cTBS treatment via accurate navigation to bilateral cerebellar dentate nucleus. Participants will be took TMS-EEG, functional magnetic resonance imaging, and diffusion tensor imaging (DTI) pre- and post- treatment. These three examinations will help to analyze the brain functional connectivity and suggest the mechanism of action of this treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged between 18 and 60,
2. Participants who are in line with the diagnostic criteria for epilepsy and drug-refractory epilepsy (DRE),
3. Participants who have duration of epilepsy ≥ 2 years and seizure frequency ≥ 2 seizures per month,
4. The type and dosage of anti-seizure medications (ASMs) keep unchanged during the experiment,
5. Participants and their families are aware of this study and sign informed consent.

Exclusion Criteria:

1. Participants who are unable to cooperate with treatment and examinations,
2. Participants who are in status epilepticus (SE),
3. Participants who are complicated with a serious infection, cerebrovascular disease, malignant tumour, and other nervous system diseases, with serious dysfunction of heart, liver, kidney, and other organs, and with psychiatric disorders,
4. Participants who are pregnant or breastfeeding,
5. Participants have contraindications of TMS and MRI, that is, the presence of metal or implanted devices in the body, such as cardiac pacemaker, deep brain stimulator, etc,
6. Participants who are in other clinical trials,
7. Participants who withdraw informed consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
TMS evoked potential amplitude change between pre- and post- treatment | 8 weeks
  TMS-EEG will be recorded pre- and post- treatment by physician and the electroencephalogram (EEG) data will be analyzed with TMS evoked potential by technician, finally, the amplitude change between pre- and post- treatment will be obtained.
functional magnetic resonance images brain functional connection change between pre- and post- treatment | 2 weeks
  Functional magnetic resonance images (fMRI) will be recorded pre- and post- treatment within 24h. Brain functional connection will be analyzed through fMRI by technician and the change of brain functional connection will be obtained.
diffusion tensor imaging fiber connectivity change between pre- and post- treatment | 12 weeks
  Diffusion tensor imaging (DTI) will be recorded pre-treatment and post-treatment in three months. DTI data will be analyzed by technician and the change of fiber connectivity change will be obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China